CLINICAL TRIAL: NCT01362504
Title: Zekai Tahir Burak Maternity Teaching Hospital Neonatal Intensive Care Unit
Brief Title: Pro-adrenomedullin as a Prognostic Marker in Neonatal Sepsis
Status: Completed | Type: Observational
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Yekta, Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: ZTB0663
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Sepsis
Keywords: Pro-adrenomedullin; Neonatal sepsis; Prognosis; Sepsis marker; Clinical sepsis; Proven sepsis
MeSH Terms: conditions — Sepsis; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Clinical sepsis
- Proven sepsis
- Control group: healthy neonates

SUMMARY:
The aim of this study was to clarify the prognostic value of serum pro-Adrenomedullin level in neonatal sepsis. Eighty term and preterm neonates with sepsis were enrolled in this study. Eighty healthy matched neonates served as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical sepsis and/or proven sepsis.

Exclusion Criteria:

* Acute kidney injury
* Intracranial hemorrhage (Grade III and IV)

Ages: 24 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm and term neonates with sepsis were enrolled in this study including 80 cases.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Neonatology Unit, Ankara, Turkey (Türkiye)